CLINICAL TRIAL: NCT02611245
Title: Phase 1 Study of NIR Fluorescence Guided Thoracic Surgery Using ICG
Brief Title: NIR Fluorescence Imaging Technique in Thoracic Surgery With ICG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Chongwei Chi, Ph.D, Assistant Professor of Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011CB707702
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer; Esophageal Cancer
Keywords: Thoracic Duct; Sentinel lymph node biopsy
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indocyanine green (Experimental): This group of patients under general anesthesia to accept conventional thoracoscopy or thoracotomy. Before systematic lymphadenectomy, four-point of ICG with 10mg was injected in normal lung tissue around the tumor. After 3-5 minutes, fluorescence and white-light images were collected and recorded in real-time. With the guidance of intraoperative images, all fluorescent lymph nodes were removed and sent to routine pathological confirmation.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — This group of patients accepted intravenous injection from 0.5mg / kg to 5mg / kg ICG within 4 to 24 hours before surgery. All patients under general anesthesia to accept conventional thoracoscopy or thoracotomy. After entering the chest using fluorescence thoracoscopy system to collect the fluorescence and white-light images and record the video. After following the routine preoperative planning surgery, the researchers will carefully assess the possibility of the benign and malignant nodules and to communicate with the families of patients. If the patient's family expressed their willingness to dissect the nodules, the researchers will remove this extra pulmonary nodules. Resected specimens will send to routine pathological confirmation compared with the fluorescence results.
  Other Names: ICG

SUMMARY:
This study aims to first apply near-infrared fluorescence imaging technology in thoracic surgery with indocyanine green in China. To evaluate the feasibility usage of the investigators' fluorescence imaging systems and the safety applications in intraoperative sentinel lymph node mapping of lung and esophageal cancer, lung nodule imaging, lung segment resection boundary determination, esophagus - tubular anastomosis, thoracic duct imaging and chylothorax repairing thoracic surgery. Aim to achieve precise boundaries definition during thoracic surgery and realize accurate, minimally invasive thoracic surgery with fluorescence imaging technology.

DETAILED DESCRIPTION:
Lung cancer is a major threat to human health. Diagnosis and treatment using precision medicine is expected to be an effective method for preventing the initiation and progression of cancer. Although anatomical and functional imaging techniques such as radiography, computed tomography (CT), magnetic resonance imaging (MRI) and positron emission tomography (PET) have played an important role for accurate preoperative diagnostics, for the most part these techniques cannot be applied intraoperatively. Optical molecular imaging is a promising technique that provides a high degree of sensitivity and specificity in tumor margin detection. Furthermore, existing clinical applications have proven that optical molecular imaging is a powerful intraoperative tool for guiding surgeons performing precision procedures, thus enabling radical resection and improved survival rates. However, detection depth limitation exists in optical molecular imaging methods and further breakthroughs from optical open surgery to minimally invasive intraoperative imaging methods are needed to develop more extensive and comprehensive intraoperative applications.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary nodules undergoing thoracoscopy or thoracotomy
* Esophageal cancer patients who underwent radical surgery
* Preoperative liver function is normal
* No indocyanine green and iodine allergies, and indocyanine green skin test negative
* Volunteered to participate in this study and signed informed consent in this study

Exclusion Criteria:

* Preoperative liver dysfunction
* Indocyanine green or iodine allergies, or indocyanine green skin test positive
* Not combined with other well-controlled comorbidities
* Clinicians considered unsuitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Detection rates of lung nodes with fluorescence imaging | 1 year
  Participants will be followed for the duration of hospital stay, an expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Chi C, Du Y, Ye J, Kou D, Qiu J, Wang J, Tian J, Chen X. Intraoperative imaging-guided cancer surgery: from current fluorescence molecular imaging methods to future multi-modality imaging technology. Theranostics. 2014 Aug 15;4(11):1072-84. doi: 10.7150/thno.9899. eCollection 2014. PMID 25250092
- [Result] Mao Y, Chi C, Yang F, Zhou J, He K, Li H, Chen X, Ye J, Wang J, Tian J. The identification of sub-centimetre nodules by near-infrared fluorescence thoracoscopic systems in pulmonary resection surgeries. Eur J Cardiothorac Surg. 2017 Dec 1;52(6):1190-1196. doi: 10.1093/ejcts/ezx207. PMID 28950327
- [Derived] Yang F, Zhou J, Li H, Yang F, Xiao R, Chi C, Tian J, Wang J. Near-infrared fluorescence-guided thoracoscopic surgical intervention for postoperative chylothorax. Interact Cardiovasc Thorac Surg. 2018 Feb 1;26(2):171-175. doi: 10.1093/icvts/ivx304. PMID 29049798
- [Derived] Li H, Zhou J, Chi C, Mao Y, Yang F, Tian J, Wang J. Clinical application of near-infrared thoracoscope with indocyanine green in video-assisted thoracoscopic bullectomy. J Thorac Dis. 2016 Jul;8(7):1841-5. doi: 10.21037/jtd.2016.06.02. PMID 27499979